CLINICAL TRIAL: NCT06159348
Title: Pilot Feasibility Study of a Novel Non-invasive Device for Diagnosis of Anemia
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Allison Judkins, Principal Investigator, University of Utah
Other Study IDs: 00145719
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Anemia
Keywords: non-invasive detection
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Participants will be adults aged 18-70, male or female
  Interventions: Diagnostic Test: Anemia Diagnostic Assistant (ADA); Diagnostic Test: Serum hemoglobin

INTERVENTIONS:
Diagnostic Test: Anemia Diagnostic Assistant (ADA) — The Anemia Diagnostic Assistant is non-invasive and simultaneously detects two markers of anemia, blood hemoglobin and the End-Tidal carbon monoxide levels. The device comprises an optical sensor module and ETCO breath sampling module.
Diagnostic Test: Serum hemoglobin — Venous blood will be drawn on the same day as the ADA was applied and sent to the hospital lab for hemoglobin analysis.

SUMMARY:
In low-resource areas of the world, anemia screening relies on analyzing a blood sample and is generally carried out in health facilities. Current anemia screening approaches have not yielded satisfactory results due to critical limitations including lack of a) reliable access to laboratory facilities, b) reliable non-invasive out-of-hospital screening tools for community health-workers, c) integration of anemia data across health systems and d) distinction between hemolytic and nutritional causes. Currently available non-invasive tools have unacceptably low accuracy and cannot distinguish between nutritional and hemolytic etiologies.

Prototype Anemia Diagnostic Assistant (ADA)

We have developed a prototype Anemia Diagnostic Assistant for non-invasive, simultaneous detection of two markers of anemia, blood hemoglobin and the End-Tidal carbon monoxide levels. The device comprises an optical sensor module and ETCO breath sampling module.

The unique and significant advantage of the instrument is its ability to detect, independently, two orthogonal variables that are required for differential diagnosis of the nutritional and hemolytic anemia:

1. Hemoglobin concentration using a non-invasive diffuse reflectance spectroscopy. Using high-fidelity, 11 wave-length spectral sensor, the device will provide optical quantification of hemoglobin levels. Optical hemoglobin sensing using diffused reflectance spectroscopy is well known, however; using traditional spectrophotometry instrumentation is very costly and thus impractical for this project. As a solution, we propose to use a validated commercially-available high accuracy 11-wavelength sensor within the visual and near-infrared (IR) range of the spectrum. The 11-wavelength spectrum will allow for sufficient accuracy in measuring the reflectance AND transmittance at isosbestic wavelengths on hemoglobin extinction curve as well as to compensate for the presence of melanin, which is a major interferant in optical determination of hemoglobin concentration. [9] The sensor was originally designed to collect data on the earlobe and/or the fingertip. Additional iterations include a sensor that straps around the wrist (similar to a smartwatch). Both versions of the device may be used in the study, and both feature standard USB or Bluetooth connectivity to ubiquitous mobile Android an iOS-based mobile platform .
2. End-tidal carbon monoxide. Using a non-invasive probe placed in proximity to the nostrils, the device will measure ETCO as a proxy measure of hemolysis. ETCO measurement as a measure for the presence of hemolysis is well documented in the medical literature and is commonly used in newborns units as a screening method for the presence of hemolysis [7,8,10]. A positive finding (presence of elevated levels of ETCO) will then prompt a referral for further hospital testing.

The objective of this study is to determine the hemoglobin and ETCO concentration in healthy volunteers using the prototype device and compare the results with the hemoglobin and ETCO concentrations obtained using standard of care devices and the CoSense system for the (ETCO measurement).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult

Exclusion Criteria:

* Immunocompromised subjects
* Patients with known hemolytic disease, anemia, or other chronic illness
* Patients who do not provide consent.
* Those who are students or reporting staff of investigators will be excluded.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from the University of Utah campus. Potential participants can be students or staff.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Difference in ADA hemoglobin values compared to serum hemoglobin values | 24 hours
  Each participant will have their hemoglobin measured using the ADA and blood analysis. These values will then be compared to measure the difference between the ADA values and the serum values.

SECONDARY OUTCOMES:
Incidence of hemolytic anemia | 24 hours
  The ETCO is a well established measure of hemolysis. The study will evaluate the number of positive readings and individual participants who have a positive measure will be referred for further hospital testing.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Judkins, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States